CLINICAL TRIAL: NCT05637762
Title: Development of a Seizure Detection Algorithm Based on Heart Rate and Movement Analysis
Acronym: DetecTeppe
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Collaborators: La Teppe Institute (Unknown)
Responsible Party: Sponsor
Other Study IDs: PLR_2022_11
Record Dates: First submitted 2022-11-08; First posted 2022-12-05 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-02

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: - EEG video recording or extension of an EEG video recording planned as part of the care - Wearing a connected heart rate and motion recording patch — The study consists of creating a database to develop an algorithm using machine learning methods.

SUMMARY:
Epilepsy is the 3rd neurological pathology after migraines and dementia syndromes with a high estimate of nearly 600,000 people affected in France. The disease is characterized by the repetition of epileptic seizures on the one hand, but also by the cognitive, behavioral, psychological and social consequences of this condition, especially when the epileptic disease is not stabilized. Epileptic patients feel a great deal of stress due to the unpredictability of the occurrence of seizures.

Seizure detection is of great interest to bioinformatics researchers and to people with epilepsy and their caregivers. Recent advances in physiological sensor technologies and artificial intelligence have opened the possibility of developing systems capable of closely monitoring the frequency of epileptic seizures with a direct impact on therapeutic adaptations. This may eventually allow for seizure prediction and/or "seizure weather" (i.e., seizure forecasting) if there is a particular chronotype of seizure occurrence for a given individual.

Currently, few devices have a sufficient level of evidence regarding their effectiveness to be recommended. Those that seem to be the most advanced are those that allow the identification of hypermotor seizures, including tonic-clonic generalized seizures and tonic-clonic secondary generalized focal seizures, mostly occurring at night. The latter represent only a small part of epileptic seizures.

The objective of the present study is to build a real life database in order to develop a seizure detection algorithm.

The recorded data will be heart rate via ECG and movement data via 9 variables measured on 3 axes x, y, z, with 3 sensors: accelerometer, gyroscope, magnetometer. These data will be collected using a connected patch available on the market (CE marking).

At the same time, the patients will benefit from a long term video-EEG examination which will be annotated by the doctors and will be used as a gold standard for the identification of seizures in order to train the algorithm.

This more complete base will be used to develop an algorithm previously developed from retrospective data.

ELIGIBILITY:
Inclusion Criteria:

* Person over 18 years of age - With drug-resistant epilepsy as defined by the International League Against Epilepsy
* Who has at least one recorded seizure with heart rate variation (i.e. tachycardia defined as an increase of 30 bpm or more than 50% over the interictal heart rate and/or bradycardia defined as a heart rate < 40 bpm or ictal asystole defined as an R-R interval greater than 3 seconds and usually lasting less than 60 seconds)
* Informed about the study and signed a consent to participate in the study (and their legal representative for patients under guardianship)
* Affiliated or beneficiary of a social insurance plan

Exclusion Criteria:

* Pregnant or breastfeeding woman
* Persons with psychogenic non-epileptic seizures (PNES)
* Person with a history of severe heart disease (myocardial infarction, heart failure, rhythm disorder, severe hypertension)
* Persons with an implantable cardiac device (pacemaker, implantable defibrillator)
* Documented allergy to hydrogel and/or acrylate
* Person benefiting from a legal protection measure other than guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The people with epilepsy will be recruited from among the patients/residents being followed for their epilepsy at the Institut La Teppe.
  Institut La Teppe is a medical and social institution that welcomes people suffering from epilepsy with cognitive deficiencies that can be severe.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2023-06-05 (Actual); Primary Completion 2025-04-24 (Actual); Study Completion 2025-04-24 (Actual)

PRIMARY OUTCOMES:
To build a training database under physiological conditions allowing the development of a detection algorithm for generalized and focal epileptic seizures in adults with epilepsy. | Day12
  Movements will be measured with accelerometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut La Teppe, Tain-l'Hermitage, France

IPD SHARING:
Plan to Share IPD: No